CLINICAL TRIAL: NCT02285465
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Multiple Oral Doses of ASP3700 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP3700 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to sponsor decision
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3700-CL-0002; 2014-003226-41 (EudraCT Number)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP3700
Keywords: Healthy volunteers; Pharmacokinetics; Pharmacodynamics; ASP3700

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP3700 multiple ascending dose cohort (Experimental)
  Interventions: Drug: ASP3700
- Placebo cohort (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP3700 — Oral
  Arms: ASP3700 multiple ascending dose cohort
Drug: Placebo — Oral
  Arms: Placebo cohort

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of ascending multiple oral doses of ASP3700 in healthy subjects.

DETAILED DESCRIPTION:
Subjects will be confined in the clinic for 18 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a skin type I, II or III (Fitzpatrick classification).
* Subject has a body mass index (BMI) of 18.5 to 30.0 kg/m2, inclusive. The subject weighs at least 50 kg at screening.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP3700 or any components of the formulation used.
* Subject does not respond to the capsaicin challenge at screening or day -1. A nonresponder is defined by a dermal blood flow (DBF) of ≤ 100% increase from baseline (normal skin) compared to DBF 30 minutes after application of 0.4 mL (approximately 300 µg) of capsaicin cream (Axsain®, 0.075% capsaicin w/w).
* Subject does not respond to the histamine challenge at screening or day -1. A nonresponder is defined by an insufficient wheal (mean diameter < 0.5 cm) and/or flare (mean diameter < 2 cm) reaction (visually assessed and measured by trained staff member) after 10 minutes of the histamine intradermal injection.
* Subject has a history of suicide attempt or suicidal behavior. Any suicidal ideation within the last 3 months (a level of 4 or 5 for any 1 item on the scale), or who are at significant risk to commit suicide, as judged by the investigator using the C-SSRS at screening and on admission to the clinical unit on day -1.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], Alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma glutamyl transferase, total bilirubin [TBL]) above the upper limit of normal (ULN). In such a case the assessment may be repeated once on day -1.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has a history of clinically significant reaction to cannabis or synthetic cannabinoids as judged by the investigator.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the investigator.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG) and protocol defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (vital sign measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) on day -1. If the mean pulse, mean SBP or mean DBP is out of the range as specified above, 1 additional triplicate measurement may be taken.
* Subject has a mean QTc(F) interval of > 430 ms (for males) and > 450 ms (for females) at day -1. If the mean QTc(F) exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject uses any prescribed or nonprescribed drugs (including antihistamines, vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day).
* Subject has used nicotine-containing products within 6 months prior to admission to the clinical unit on day -1.
* Subject has a history of drinking > 21 units of alcohol per week for male subjects or > 14 units of alcohol for female subjects (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit on day -1.
* Subject has used any drugs of abuse within 3 months prior to admission to the clinical unit on day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit on day -1.
* Subject has consumed grapefruit, grapefruit-containing products, Seville orange-containing products, caffeine, xanthine, quinidine or theobromine containing products within 72 hours prior to admission to the clinical unit on day -1.
* Subject has had a significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit on day -1.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (antiHAV [IgM]), hepatitis C virus antibodies (antiHCV), or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject has participated in any clinical study or has been treated with any investigational drugs within 3 months or 5 half-lives, whichever is longer, prior to screening.
* Subject has a skin disease, acute or chronic (e.g., atopic dermatitis) or any active dermatological conditions, local pigmentary disorders, or body art (e.g., tattoos) that might interfere with the clinical study assessments.
* Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for clinical study participation.
* Subject is an employee of the Astellas Group or Contract Research Organization (CRO) involved in the clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | up to end of study visit (up to 26 days)
Safety as assessed by vital signs | up to end of study visit (up to 26 days)
Safety as assessed by orthostatic evaluation | Days 1 and 14
Safety as assessed by laboratory tests | up to end of study visit (up to 26 days)
  Laboratory tests include hematology, biochemistry and urinalysis.

SECONDARY OUTCOMES:
Safety profile: Routine 12-lead ECG, C-SSRS, ARCI-49, Bond and Lader VAS, continuous cardiac monitoring (12-lead Holter ECG), exploratory sex hormone-related and renal biomarkers | up to end of study visit (up to 26 days)
  Electrocardiogram (ECG); Columbia-Suicide Severity Rating Scale (C-SSRS); Addiction Research Center Inventory(ARCI)-49 (49-item); Visual Analog Scale (VAS).
Pharmacokinetics profile of ASP3700 (plasma): Cmax, tmax, tlag | Cmax, tmax = Days 1 and 14; tlag = Day 1
  Maximum concentration (Cmax); time of maximum concentration (tmax); time prior to the time corresponding to the first measurable (nonzero) concentration (tlag)
Pharmacokinetics profile of ASP3700 (plasma): AUCtau, CL/F, λz, MRT, t1/2, Vz/F, Rac (AUC), Rac (Cmax), PTR | Day 14
  Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau); apparent oral clearance (CL/F); terminal elimination rate constant (λz); mean residence time (MRT); terminal elimination half-life (t1/2); apparent volume of distribution during terminal elimination phase after extravascular dosing (Vz/F); accumulation ratio based on AUE (Rac[AUC]); accumulation ratio based on Cmax (Rac[Cmax]); peak-trough ration (PTR)
Pharmacokinetics parameter of ASP3700 (plasma): Ctrough | Days 4, 6, 8, 10, 14 and 15
  Concentration immediately prior to dosing at multiple dosing (Ctrough)
Pharmacokinetics profile of ASP3700 (urine): Ae24, Ae24%, Aetau, Aetau% | Ae24, Ae24% = Day 1; Aetau, Aetau% = Day14
  Cumulative amount of drug excreted in the urine from Time Zero to 24 hours (Ae24); percent fraction of administered drug excreted unchanged in the urine from time zero to 24 hours (Ae24%); cumulative amount of drug excreted in the urine over the dosing interval at steady-state (Aetau); percent fraction of administered drug excreted unchanged in the urine over the dosing interval at steady-state (Aetau%)
Pharmacokinetics parameter of ASP3700 (urine): CLR | Days 1 and 14
  Renal clearance (CLR)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.